CLINICAL TRIAL: NCT00826423
Title: Pilot Study to Assess Safety and Efficacy of Short Course Multiple Drug Therapy for Adult Patients With Mycobacterium Avium Intracellulare Complex (MAC) Infection Associated With Mulit Focal Bronchiectasis and Multiple Small Nodules
Brief Title: Mycobacterium Avium Intracellulare Complex (MAC) Study
Acronym: MAC
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Dr. Jack P. Leventhal, Mayo Clinic
Other Study IDs: 07-004414
Record Dates: First submitted 2009-01-20; First posted 2009-01-22 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-07

CONDITIONS: Mycobacterium Avium Intracellulare Complex (MAC)
Keywords: treatment with Triple antibiotic therapy
MeSH Terms: conditions — Mycobacterium avium-intracellulare Infection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — sputum and blood collection for analysis
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is short course (3 month) multiple drug antibiotic therapy. The purpose of this research study is to evaluate the clinical and radiology response to assess whether drug resistance develops and assess quality of life measures with MAC disease.

DETAILED DESCRIPTION:
The goal of this pilot study is to assess the safety and efficacy of short course (3 months) multiple drug antimicrobial therapy in adults with MAC pulmonary disease associated with multifocal bronchiectasis and multiple small nodules. We propose to evaluate the clinical and radiographic response, assess whether macrolide (either Clarithromycin or Azithromycin) resistance develops, and assess quality of life measures.

No evidence of efficacy is required to proceed to longer term studies; however, we will need to confirm lack of development of macrolide resistance in this pilot study before proceeding to any additional studies to evaluate the efficacy of short course MAC treatment.

Once we have demonstrated the feasibility of short course therapy and confirm that resistance to macrolides does not develop, we hope to apply for external funding to support a longer term randomized controlled trial comparing "standard" MAC therapy (which usually consists of a period of eighteen to twenty-four months with at least three antimicrobials) to short course (three months) MAC antimicrobial treatment, alternating each year with nine months of non-MAC bronchial hygiene measures for two consecutive years. If a larger study confirms efficacy of this approach, we would then propose even larger multi-site studies to test the hypothesis that short course MAC therapy alternating every year with non-MAC bronchial hygiene therapy should be considered in all adult patients with MAC pulmonary disease associated with multifocal bronchiectasis and multiple small nodules throughout their lives.

The longer term goal of this research is to develop an optimal treatment strategy for these patients (in whom MAC will likely persist indefinitely) that will result in not only a better quality of life, but less evidence of long term lung damage, less risk of drug-related morbidity, and be better tolerated by the patients compared to current treatment strategies.

The specific aims of this pilot study are as follows:

Primary Aim:

1. Confirm that macrolide (either Clarithromycin or Azithromycin) resistance does not develop as a result of short course treatment.

   Secondary Aims:
2. Assess for change in quality of life metrics (St. George Respiratory Questionnaire and SF 12) from baseline to the conclusion of the study period (six months). We expect to see improvement in quality of life measures as a result of this short course treatment trial.
3. Assess for change in pulmonary function from baseline to the conclusion of the study period. We expect to see improvement particularly in the FEV1, FEV1/FVC, and diffusing capacity for carbon monoxide as a result of this short course treatment trial.
4. Assess for change in high resolution computerized tomography (HRCT) of the chest, evidence of MAC pulmonary disease (multifocal bronchiectasis associated with multiple small nodules) from baseline to the conclusion of the study period. We do not anticipate being able to demonstrate improvement in the HRCT evidence of MAC lung disease during the short period of this trial since these changes usually occur quite slowly.

ELIGIBILITY:
Inclusion Criteria:

1. All patients must meet diagnostic criteria for nontuberculous mycobacterial pulmonary disease as per ATS/IDSA Official Statement (AJRCCM Vol 175 pp 367-416, 2007)
2. Confirmation both by a chest radiologist and the investigators of multifocal bronchiectasis and multiple small nodules on HRCT scanning of the chest
3. Repeatedly positive sputum cultures and/or bronchial washings for MAC (in accordance with microbiologic diagnostic criteria outline by the American Thoracic Society)
4. MAC must be proven to be macrolide (either Clarithromycin or Azithromycin) sensitive at the onset of the study
5. Age greater than 18
6. No active treatment for MAC lung disease within the past two years
7. Patients and their physicians must be willing to discontinue other non-MAC antimicrobials which may have been used as part of their pre-study bronchial hygiene program.

Exclusion Criteria:

1. History of Cystic Fibrosis or HIV disease
2. Known allergy or intolerance to any of the proposed antibiotics
3. Inability to return at three month intervals for testing over the six month study period
4. Inability to complete quality of life questionnaires
5. Pregnancy
6. Presence of any abnormality on baseline ophthalmological examination which would preclude the use of ethambutol.
7. Coexistence of non-tuberculous mycobacteria other than MAC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Fifteen adult patients will be included in this pilot study. This sample size was chosen not on the basis of formal statistical considerations. However, data from 15 patients will be sufficient to provide rough preliminary estimates of parameters that may be needed for developing power statements for a follow-up larger (randomized) trial. If macrolide resistance occurs in 5% or less of patients in this population, with ≥83% probability only one or zero of the 15 patients will develop resistance. If two or more of the 15 patients develop resistance then further investigations of resistance will be warranted before moving on to randomized trials.
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2008-06; Primary Completion 2011-06 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jack P Leventhal, MD, Principal Investigator — Mayo Clinic Assistant Professor of Medicine
Locations (1):
- Mayo Clinic, Jacksonville, Florida, United States